CLINICAL TRIAL: NCT06405750
Title: Left Atrial Appendage Arrhythmogenic and Thrombogenic Substrate
Acronym: LAATAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Helena DOMINGUEZ, MD, PhD, Associate Professor, University Hospital Bispebjerg and Frederiksberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-23015282; P-2023-227 (Other: Capital Region Denmark)
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: heart surgery; atrial myocardiopathy; arrhythmogenic substrate; stroke; cerebral transitory ischemic attack; thrombogenesis; cardiac embolism
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Intervention Model Description: Mechanistic study based on analysis of biological material collected along with electrocardiogram features on individuals undergoing open-heart surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LAA closure (Other): All patients included in the study undergo closure of the Left Atrial Appendage
  Interventions: Procedure: left atrial appendage closure

INTERVENTIONS:
Procedure: left atrial appendage closure — systematic closure of the left atrial appendage in addition to the planned heart surgery

SUMMARY:
The purpose of the project is to elucidate whether it is possible to identify which patients are at risk of forming blood clots that can cause stroke based on analysis of the electrocardiogram.

In connection with the operation, the small pouch known as the auricle of the heart is closed, which can be completely removed after closing. This procedure is common in patients with atrial fibrillation to protect the brain from stroke. In the project, all patients will have this auricle closed if they agree to participate in the project.

After closure, the auricle is usually discarded. We will analyze the blood and the auricle tissue taken (if available) in connection with the operation itself, together with the analysis of the electrocardiogram recorded before the planned heart operation.

DETAILED DESCRIPTION:
Patients scheduled for elective heart surgery are invited to participate. After informed consent is signed, an ECG and blood samples are gathered the day before surgery or the same day of the surgery is planned.

During surgery, the patients undergo closure of the left atrial appendage (LAA). The choice of the device is at the discretion of the surgeon. If possible, the entire LAA is removed and processed for further analysis. The right atrial appendage is likewise removed and follows the same procedure as the LAA.

The analyses include measurement of up-/down-regulated thrombosis factors and inflammatory markers.

The right and left atrial appendage tissue collected are immediately processed for micro-patch-clamp studies, and the remaining tissue is divided into a part that is frozen for later analyses and a part that is fixed and embedded in paraffin for further histological analyses.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent AND
* planned any open-heart surgery:

  * CABG
  * valve repair or replacement
  * aorta surgery
  * any combination of the above

Exclusion Criteria:

* current endocarditis
* follow-up not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
stroke | six years
  number of patients with clinical stroke

SECONDARY OUTCOMES:
perioperative atrial fibrillation | 30 days
  number of patients with incident atrial fibrillation the days after surgery, prior to discharge
silent brain infarctions | six years
  number of patients in whom asymptomatic ischemic infarctions are identified in brain scans (CTC or MRI)
occurrence of atrial fibrillation during follow-up | ten years

CONTACTS AND LOCATIONS:
Overall Officials: Helena Dominguez, Study Director — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Rigshospitalet, Copenhagen, Denmark